CLINICAL TRIAL: NCT03580720
Title: Diaphragm Electromyography to Estimate Breathing Effort: a Physiological Study
Brief Title: Electromyography for Diaphragm Effort
Acronym: Edi2Pdi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof.dr. L.M.A. Heunks, Clinical professor, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL64648.029.18
Record Dates: First submitted 2018-06-08; First posted 2018-07-09 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Diaphragm Injury; Muscle Weakness; Weaning Failure; Physiological Stress
Keywords: Monitoring; Breathing effort; Intensive Care; Diaphragm weakness
MeSH Terms: conditions — Muscle Weakness; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intervention group, receiving Inspiratory threshold loading protocol.
  Interventions: Other: Inspiratory threshold loading protocol

INTERVENTIONS:
Other: Inspiratory threshold loading protocol — Subjects will be instrumented with catheters that measure electrical activity of the diaphragm and transdiaphragmatic pressure. Subjects will perform a stepwise inspiratory threshold loading protocol to induce a wide range of diaphragm activity.

SUMMARY:
Mechanical ventilation may be necessary to save the life of a patient due to an accident, pneumonia or surgery. The ventilator then temporarily takes over the function of the respiratory muscles. During treatment in the Intensive Care, the amount of support provided by the ventilator is usually lowered gradually, until the point that the patient can breathe unassisted once again. However, in a large fraction of patients (up to 40%) it takes days to weeks before the patient is able to breathe unassisted, even after the initial disease has been treated. This is called prolonged weaning.

A possible cause of prolonged weaning is weakness of the respiratory muscles. The diaphragm, the largest respiratory muscle, can become weakened if it is used too little, much like all other muscles in the body. Additionally, damage and weakness of the diaphragm can occur when the diaphragm has to work excessively. Therefore, it is important that the diaphragm works enough; not so little that it becomes weakened, but not too much either.

Measurements of pressure generated by the diaphragm are needed to determine the current level of diaphragm activity in a patient on mechanical ventilation. However, these measurements are rarely performed, because they are time-consuming and require placement of two additional nasogastric catheters. This is a shame, as adequate loading of the diaphragm might prevent development of weakness, leading to shorter duration of mechanical ventilation. Finding alternative measurements of diaphragm effort might be a solution to this problem.

It has been hypothesized that the electrical activity of the diaphragm provides a reliable indication of diaphragm effort. This study aims to determine whether there is a correlation between pressure generation by the diaphragm and electrical activity of the diaphragm over a wide range of respiratory activity, from low effort to extreme effort, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Age >18 years

Exclusion Criteria:

* History of cardiac and/or pulmonary disease or current medication use
* History of pneumothorax
* Contra-indications for nasogastric tube placement (recent epistaxis, severe coagulopathy, current upper airway pathology)
* Contra-indication for magnetic stimulation (cardiac pacemakers or metal in cervical area)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Electrical activity of the diaphragm | Electrical activity of the diaphragm will be assessed at multiple levels of breathing effort in each subject for two hours.
  Diaphragm electromyography will be obtained with multiple electrode pairs situated on specialized esophageal catheters. The raw diaphragm electromyography will be filtered and integrated to obtain the compound mean action potential reported in microvolts (μV) as described in ref 1 (Sinderby et al.).
Transdiaphragmatic pressure | Transdiaphragmatic pressure will be assessed at multiple levels of breathing effort in each subject for two hours.
  The pressure gradient over the diaphragm will be obtained by subtracting the esophageal pressure from the pressure in the stomach, measured with specialized catheters, and will be reported in centimeters of water (cmH2O) as described in ref 3, American Thoracic Society (ATS) statement on respiratory muscle testing.

SECONDARY OUTCOMES:
Work of breathing | Work of breathing will be assessed at multiple levels of breathing effort in each subject for two hours.
  Work of breathing will be obtained by integrating the pressure-volume loops of esophageal pressure and tidal volume, and will be reported in Joule per minute as described in ref 3, ATS statement on respiratory muscle testing..
Pressure-time product of the diaphragm | Pressure-time product of the diaphragm will be assessed at multiple levels of breathing effort in each subject for two hours.
  Pressure-time product of the diaphragm will be obtained by dividing the time-integral of transdiaphragmatic pressure (described above) over time, and will be reported as cmH20*s per minute as described in ref 3, ATS statement on respiratory muscle testing..
Pressure-time product of the respiratory muscles | Pressure-time product of the respiratory muscles will be assessed at multiple levels of breathing effort in each subject for two hours.
  Pressure-time product of the respiratory muscles will be obtained by dividing the time-integral of esophageal pressure over time, and will be reported as cmH20*s per minute as described in ref 3, ATS statement on respiratory muscle testing..
Mechanical power | Mechanical power will be assessed at multiple levels of breathing effort in each subject for two hours.
  Mechanical power will be obtained by multiplying the work of breathing (described above) by the number of breaths per minute, and will be reported in Watt (joule/minute) as described in ref 3, ATS statement on respiratory muscle testing..

OTHER OUTCOMES:
Accessory muscle recruitment | Two hours.
  As an explorative end-point, the timepoint at which several accessory inspiratory muscles are recruited during incremental respiratory loading will be studied and reported (if technically possible)
Diaphragm thickening fraction. | Thickening fractions will be obtained at multiple levels of breathing effort in each subject for up to two hours
  Using a linear probe positioned in the mid-axillary line the diaphragm will be visualized as per clinical protocol. Diaphragm thickness will be measured during inspiration and expiration and will be reported in mm. Thickening fraction will be obtained with the following formula: (Thickness during inspiration - thickness during expiration) / thickness during expiration * 100% as described in ref 2 (Vivier et al.).

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Spoelstra - de Man, MD, PhD, Study Chair — Amsterdam UMC, location VUmc; Leo Heunks, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sinderby CA, Beck JC, Lindstrom LH, Grassino AE. Enhancement of signal quality in esophageal recordings of diaphragm EMG. J Appl Physiol (1985). 1997 Apr;82(4):1370-7. doi: 10.1152/jappl.1997.82.4.1370. PMID 9104877
- [Background] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831